CLINICAL TRIAL: NCT03797313
Title: Observational Study of Expected Acute Respiratory Failure (ARF) Recovery
Brief Title: Observational Study of Expected ARF Recovery
Acronym: OSEAR
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00197235; 00181895 (Other: Other); K01HL141637-01 (NIH)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-02

CONDITIONS: Acute Respiratory Failure; Post Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient's expectations met at Hospital discharge: ARF survivors whose expectations for recovery at hospital discharge are fully met 6 months later.
- Patient's with unmet expectations at Hospital Discharge: ARF survivors whose expectations for recovery at hospital discharge are not fully met 6 months later.

SUMMARY:
This is an observational cohort study of the association between patient expectations for functional recovery and quality of life among acute respiratory failure survivors 6 months after hospital discharge.

DETAILED DESCRIPTION:
This study will enroll adults who are diagnosed with acute respiratory failure during an ICU admission and discharged from the ICU alive. All participants will receive usual clinical care. Participant expectations for functional recovery will be assessed before hospital discharge via a standardized questionnaire containing a visual analogue scale and questions about expected ability and importance of being able to perform activities of daily living and instrumental activities of daily living in 6 months. At 6 months, participants will be re-contacted by phone. Study staff will administer questionnaires to assess whether patient expectations have been met. Quality of life will be assessed using the WHOQOL-BREF and the EQ-5D-VAS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Respiratory failure managed in the ICU, where respiratory failure is defined as ≥1 of the following:
* Mechanical ventilation via an endotracheal tube ≥ 24 hours OR
* Non-invasive ventilation (CPAP, BiPAP) ≥ 24 consecutive hours* provided for acute respiratory failure (not for Obstructive Sleep Apnea or other stable use) OR
* High flow nasal cannula with FIO2 ≥ 0.5 and flow rate ≥ 30 LPM for ≥ 24 consecutive hours*

  *Occasional rest periods of ≤ 1 hour each are not deducted from the calculation of consecutive hours.
* Expected by the clinical team to be discharged home alive

Exclusion Criteria:

* Patient in ICU < 24 hours
* Mechanical ventilation at baseline or mechanical ventilation solely for airway protection or obstruction
* Residing in a medical institution at the time of hospital admission
* Homeless / Prisoner / Primary residence not in the USA / Unable to communicate by telephone in English
* More than mild dementia (either known diagnosis of moderate or worse dementia or IQ-CODE > 3.6; screening performed on patients > 50 years old or with family reports of possible memory decline)
* Patient on hospice at or before time of enrollment
* Patients who, based solely on pre-existing medical problems (such as poorly controlled neoplasm or other end stage disease, including Stage IV heart failure or severe burns), would not be expected to survive 6 months in the absence of the acute respiratory failure.
* Patients with neurological injury either receiving treatment for intracranial hypertension or who are not expected to return to consciousness.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: survivors of acute respiratory failure (ARF) who are expected to be discharged home alive.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of life measured using the World Health Organization Quality of Life-BREF instrument (WHOQOL-BREF) after hospital discharge | 6 months after hospital discharge
  WHOQOL-BREF is a measure of overall quality of life that evaluates satisfaction with important aspects of life rather than of health. The instrument contains 26 items across 4 domains, and requires approximately 5 minutes to administer over the phone. The 26 items in the WHOQOL-BREF are scored in four domains: physical, psychological, social relations, and environment, with between 3 and 8 items in each domain and two "benchmark" items addressing overall QoL. Transforming the raw scores results in a domain score between 0 - 100, enabling comparisons between domains with different numbers of items. Higher scores indicate greater participant satisfaction with their quality of life and lower scores indicate worse satisfaction with quality of life.

SECONDARY OUTCOMES:
Patient expectation error measure using EQ-5D VAS | 6 months after hospital discharge
  A secondary analysis will estimate patient expectation error, defined as the difference between the health-related quality of life score expected at hospital discharge and the actual health related quality of life score assessed using the EQ-5D VAS 6 months after hospital discharge. The EQ-5D VAS ranges from 0 to 100 with 0 representing the worst imaginable health state and 100 representing the best imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Turnbull, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Vanderbilt University, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Cox CE, Docherty SL, Brandon DH, Whaley C, Attix DK, Clay AS, Dore DV, Hough CL, White DB, Tulsky JA. Surviving critical illness: acute respiratory distress syndrome as experienced by patients and their caregivers. Crit Care Med. 2009 Oct;37(10):2702-8. doi: 10.1097/CCM.0b013e3181b6f64a. PMID 19865004
- [Background] Spragg RG, Bernard GR, Checkley W, Curtis JR, Gajic O, Guyatt G, Hall J, Israel E, Jain M, Needham DM, Randolph AG, Rubenfeld GD, Schoenfeld D, Thompson BT, Ware LB, Young D, Harabin AL. Beyond mortality: future clinical research in acute lung injury. Am J Respir Crit Care Med. 2010 May 15;181(10):1121-7. doi: 10.1164/rccm.201001-0024WS. Epub 2010 Mar 11. PMID 20224063
- [Background] Zambon M, Vincent JL. Mortality rates for patients with acute lung injury/ARDS have decreased over time. Chest. 2008 May;133(5):1120-7. doi: 10.1378/chest.07-2134. Epub 2008 Feb 8. PMID 18263687
- [Background] Phua J, Badia JR, Adhikari NK, Friedrich JO, Fowler RA, Singh JM, Scales DC, Stather DR, Li A, Jones A, Gattas DJ, Hallett D, Tomlinson G, Stewart TE, Ferguson ND. Has mortality from acute respiratory distress syndrome decreased over time?: A systematic review. Am J Respir Crit Care Med. 2009 Feb 1;179(3):220-7. doi: 10.1164/rccm.200805-722OC. Epub 2008 Nov 14. PMID 19011152
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Hopkins RO, Suchyta MR, Kamdar BB, Darowski E, Jackson JC, Needham DM. Instrumental Activities of Daily Living after Critical Illness: A Systematic Review. Ann Am Thorac Soc. 2017 Aug;14(8):1332-1343. doi: 10.1513/AnnalsATS.201701-059SR. PMID 28463657
- [Background] Kamdar BB, Huang M, Dinglas VD, Colantuoni E, von Wachter TM, Hopkins RO, Needham DM; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Network. Joblessness and Lost Earnings after Acute Respiratory Distress Syndrome in a 1-Year National Multicenter Study. Am J Respir Crit Care Med. 2017 Oct 15;196(8):1012-1020. doi: 10.1164/rccm.201611-2327OC. PMID 28448162
- [Background] Lieu TA, Au D, Krishnan JA, Moss M, Selker H, Harabin A, Taggart V, Connors A; Comparative Effectiveness Research in Lung Diseases Workshop Panel. Comparative effectiveness research in lung diseases and sleep disorders: recommendations from the National Heart, Lung, and Blood Institute workshop. Am J Respir Crit Care Med. 2011 Oct 1;184(7):848-56. doi: 10.1164/rccm.201104-0634WS. PMID 21965016
- [Background] Carson SS, Goss CH, Patel SR, Anzueto A, Au DH, Elborn S, Gerald JK, Gerald LB, Kahn JM, Malhotra A, Mularski RA, Riekert KA, Rubenfeld GD, Weaver TE, Krishnan JA; American Thoracic Society Comparative Effectiveness Research Working Group. An official American Thoracic Society research statement: comparative effectiveness research in pulmonary, critical care, and sleep medicine. Am J Respir Crit Care Med. 2013 Nov 15;188(10):1253-61. doi: 10.1164/rccm.201310-1790ST. PMID 24160906
- [Background] Cox CE, Martinu T, Sathy SJ, Clay AS, Chia J, Gray AL, Olsen MK, Govert JA, Carson SS, Tulsky JA. Expectations and outcomes of prolonged mechanical ventilation. Crit Care Med. 2009 Nov;37(11):2888-94; quiz 2904. doi: 10.1097/CCM.0b013e3181ab86ed. PMID 19770733
- [Background] Lamas DJ, Owens RL, Nace RN, Massaro AF, Pertsch NJ, Gass J, Bernacki RE, Block SD. Opening the Door: The Experience of Chronic Critical Illness in a Long-Term Acute Care Hospital. Crit Care Med. 2017 Apr;45(4):e357-e362. doi: 10.1097/CCM.0000000000002094. PMID 27632675
- [Background] Turnbull AE, Davis WE, Needham DM, White DB, Eakin MN. Intensivist-reported Facilitators and Barriers to Discussing Post-Discharge Outcomes with Intensive Care Unit Surrogates. A Qualitative Study. Ann Am Thorac Soc. 2016 Sep;13(9):1546-52. doi: 10.1513/AnnalsATS.201603-212OC. PMID 27294981
- [Background] Thompson AG, Sunol R. Expectations as determinants of patient satisfaction: concepts, theory and evidence. Int J Qual Health Care. 1995 Jun;7(2):127-41. doi: 10.1093/intqhc/7.2.127. PMID 7655809
- [Background] Gonzalez Saenz de Tejada M, Escobar A, Herrera C, Garcia L, Aizpuru F, Sarasqueta C. Patient expectations and health-related quality of life outcomes following total joint replacement. Value Health. 2010 Jun-Jul;13(4):447-54. doi: 10.1111/j.1524-4733.2009.00685.x. Epub 2010 Jan 15. PMID 20088892
- [Background] Soroceanu A, Ching A, Abdu W, McGuire K. Relationship between preoperative expectations, satisfaction, and functional outcomes in patients undergoing lumbar and cervical spine surgery: a multicenter study. Spine (Phila Pa 1976). 2012 Jan 15;37(2):E103-8. doi: 10.1097/BRS.0b013e3182245c1f. PMID 21629159
- [Background] Hamilton DF, Lane JV, Gaston P, Patton JT, Macdonald D, Simpson AH, Howie CR. What determines patient satisfaction with surgery? A prospective cohort study of 4709 patients following total joint replacement. BMJ Open. 2013 Apr 9;3(4):e002525. doi: 10.1136/bmjopen-2012-002525. Print 2013. PMID 23575998
- [Background] Pihl K, Roos EM, Nissen N, JoRgensen U, Schjerning J, Thorlund JB. Over-optimistic patient expectations of recovery and leisure activities after arthroscopic meniscus surgery. Acta Orthop. 2016 Dec;87(6):615-621. doi: 10.1080/17453674.2016.1228411. Epub 2016 Sep 13. PMID 27622598
- [Background] Waljee J, McGlinn EP, Sears ED, Chung KC. Patient expectations and patient-reported outcomes in surgery: a systematic review. Surgery. 2014 May;155(5):799-808. doi: 10.1016/j.surg.2013.12.015. Epub 2013 Dec 16. PMID 24787107
- [Background] Aversa M, Chowdhury NA, Tomlinson G, Singer LG. Preoperative expectations for health-related quality of life after lung transplant. Clin Transplant. 2018 Oct;32(10):e13394. doi: 10.1111/ctr.13394. Epub 2018 Sep 25. PMID 30160803
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Charney DS. Psychobiological mechanisms of resilience and vulnerability: implications for successful adaptation to extreme stress. Am J Psychiatry. 2004 Feb;161(2):195-216. doi: 10.1176/appi.ajp.161.2.195. PMID 14754765
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Cosco TD, Kaushal A, Richards M, Kuh D, Stafford M. Resilience measurement in later life: a systematic review and psychometric analysis. Health Qual Life Outcomes. 2016 Jan 28;14:16. doi: 10.1186/s12955-016-0418-6. PMID 26821587
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Shumaker SC, Frazier SK, Moser DK, Chung ML. Psychometric Properties of the Multidimensional Scale of Perceived Social Support in Patients With Heart Failure. J Nurs Meas. 2017 Apr 1;25(1):90-102. doi: 10.1891/1061-3749.25.1.90. PMID 28395702
- [Background] Hoffmann TC, Del Mar C. Patients' expectations of the benefits and harms of treatments, screening, and tests: a systematic review. JAMA Intern Med. 2015 Feb;175(2):274-86. doi: 10.1001/jamainternmed.2014.6016. PMID 25531451
- [Derived] Turnbull AE, Lee EM, Dinglas VD, Beesley S, Bose S, Banner-Goodspeed V, Hopkins RO, Jackson JC, Mir-Kasimov M, Sevin CM, Brown SM, Needham DM; APICS-01 Study Team. Fulfillment of Patient Expectations after Acute Respiratory Failure: A Multicenter Prospective Cohort Study. Ann Am Thorac Soc. 2023 Apr;20(4):566-573. doi: 10.1513/AnnalsATS.202207-600OC. PMID 36227771